# Treatment-Resistant Depression Augmentation Therapy with An Analog of the Neuroactive Steroid Allopregnanolone: A Pilot Study

NCT02900092

Version Date: 11/8/18

### I. BIOSTATISTICAL ANALYSIS

## A. Specific data variables being collected for the study (e.g., data collection sheets)

**Table 1. Schedule of Clinician and Patient** 

**Ratings** 

| Clinician<br>Rating | Screening | Baseline | Week<br>2 | Week<br>4 | Week<br>6 | Week<br>8 | Week<br>10 | 3 Mo<br>Follow<br>up |
|---|---|---|---|---|---|---|---|---|
| SCID and MGH | | | | | | | | |
| ATRQ | Х | | | | | | | |
| MADRS | Х | X | X | Х | Х | Х | Х | |
| CGI-I, S | | X | X | Х | Х | Х | Х | |
| HAM-D | | Х | | | | Х | | |
| Patient | | | | | | | | |
| Rating | | | | | | | | |
| SDQ | | Х | Х | Х | Х | Х | Х | Х |
| IDS-SR | | X | X | Х | Х | Х | Х | Х |
| SF-36 | | X | X | Х | Х | Х | Х | |
| CHRT | | X | X | Х | Х | X | Х | |
| SAFTEE-SI | | X | X | Х | Х | X | Х | |
| CPFQ | | X | X | Х | Х | X | Х | |
| BFI | | X | Χ | Х | Х | Х | Х | Х |
| ESS | | X | Χ | Х | Х | Х | Х | |
| FSS | | X | Χ | Х | Х | Х | Х | |
| DISF | | X | X | Х | Х | Χ | Х | |
| SFQ | | X | X | Х | Х | Х | Х | |
| GAD-7 | | X | Χ | Х | Х | Х | Х | Х |
| Probabilistic | | | | | | | | |
| Reward | | | | | | | х | |
| Task | | X | | | | | | |
| Pattern | | | | | | | | |
| Separation | | | | | | | Х | |
| Task | | X | | | | | | |

### **B. Study Endpoints**

The primary endpoint will be change in depression severity as measured by the change in MADRS from baseline to 8 weeks. Secondary endpoints of efficacy include both self-rated and clinician-rated assessments as listed below.

## C. Statistical Methods

Data will be examined for normality using Shapiro-Wilk testing and log-transformed if not normally distributed. Longitudinal data will be analyzed using paired T tests. Univariate regression modeling will be performed to determine whether an increase in allopregnanolone levels predict an improvement in depression symptom severity. **Power Analysis** 

**Determination of an n=10 women with treatment-resistant depression:** Based on our pilot data of the effect of low-dose testosterone on depresion severity in nine women with treatment-resistant depression in which there was an effect size of 10.7 points on the MADRS with an SD 7.5, we will have ample power to detect a clinically significant effect size with the proposed sample size.<sup>13</sup> The data from this study will provide an effect size for power calculations for applications for further funding.